CLINICAL TRIAL: NCT01486602
Title: Phase I Study of Accelerated Hypofractionated Radiation Therapy With Concomitant Chemotherapy for Unresectable Stage III Non-Small Cell Lung Cancer
Brief Title: Specialized Radiation Therapy and Chemotherapy in Treating Patients With Stage III Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB 31102; CDR0000719011 (Registry Identifier: Physician Data Query); NCI-2012-00087 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA031946 (NIH); U10CA180821 (NIH)
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Concurrent therapy + consolidation therapy (Experimental): Concurrent Therapy (1 cycle = 14 days, Cycles 1-3): Patients will receive paclitaxel 45 mg/m^2 by IV over 1 hour weekly followed by carboplatin AUC 2 by IV over 30-60 minutes for 4 weeks (there will be no chemotherapy during Cycle 3). Patients will receive radiotherapy concurrently for up to 5.5 weeks, depending on the cohorts the patient is registered defined per the protocol.
  Consolidation Therapy (1 cycle = 21 days, Cycles 4-5): Four weeks following the end of radiotherapy patients will receive paclitaxel 200 mg/m^2 by IV over 3 hours followed by carboplatin AUC 6 by IV over 30-60 minutes on day 1 of each 21 day cycle for a total of 2 cycles (days 1 and 22).
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — IV
Drug: paclitaxel — IV
Radiation: radiation therapy — Defined per the protocol

SUMMARY:
This phase I trial studies the side effects and the best dose of hypofractionated radiation therapy when given together with chemotherapy in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving hypofractionated radiation therapy together with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerable radiotherapy (RT) dose fraction for accelerated hypofractionated radiotherapy with concurrent chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the rate of radiographic response to treatment. II. To estimate the rates of progression: local/regional/distant. III. To estimate the progression-free survival. IV. To estimate the overall survival.

OUTLINE: This is a dose-escalation study of accelerated hypofractionated radiotherapy.

CONCURRENT THERAPY: Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30-60 minutes on days 1 and 8. Treatment repeats every 14 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo accelerated hypofractionated radiotherapy using 3-dimensional conformal radiation therapy or intensity-modulated radiotherapy (IMRT) once daily, 5 days a week, for approximately 4-5.5 weeks.

CONSOLIDATION THERAPY: Beginning 4 weeks after completion of radiotherapy, patients receive paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
1. Histologically or cytologically documented non-small cell lung cancer
2. Stage IIIA or IIIB non-small cell lung cancer (NSCLC) per American Joint Committee on Cancer (AJCC) version 7; patients who present with N2 or N3 disease and an undetectable primary tumor are also eligible
3. Thoracic disease without supraclavicular or contralateral hilar involvement
4. When pleural fluid is visible on both computed tomography (CT) scan and on a chest x-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative; exudative pleural effusions are excluded regardless of cytology; patients with effusions that are minimal (i.e., not visible on chest x-ray) and too small to safely tap are eligible
5. No prior radiotherapy or chemotherapy for NSCLC
6. No prior mediastinal or thoracic radiotherapy
7. Patients with complete surgical resection of disease are not eligible, however; patients with surgical resection and measurable gross residual disease present on imaging are considered eligible
8. Patients must have measurable disease

   * Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2 cm with conventional techniques or as >= 1 cm with spiral CT scan
   * Patients with non-measurable disease are not eligible; all other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly nonmeasurable lesions; lesions that are considered non-measurable include the following:

     * Bone lesions
     * Leptomeningeal disease
     * Ascites
     * Pleural/pericardial effusion
     * Inflammatory breast disease
     * Lymphangitis cutis/pulmonis
     * Abdominal masses that are not confirmed and followed by imaging techniques
     * Cystic lesions
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
10. No patients that are known to be pregnant or nursing
11. Granulocytes ≥ 1,500/μl Platelet count ≥ 100,000/μl Bilirubin ≤ 1.5 times upper limit of normal (ULN) Aspartate aminotransferase (AST) (serum glutamic oxalo-acetic transaminase [SGOT]) ≤ 2.0 times ULN Serum creatinine ≤ 1.5 times ULN OR calculated creatinine clearance >= 70 mL/min FEV-1 ≥ 1.2 L/sec or 50% predicted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated RT dose fraction | Up to 28 months

SECONDARY OUTCOMES:
Radiographic response | Up to 5 years
Metabolic response | Up to 5 years
Rates of progression: local/regional/distant | Up to 5 years
Progression-free survival | Up to 5 years
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: James J. Urbanic, MD, Study Chair — Wake Forest University Health Sciences
Locations (11):
- United States (11):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Moores University of California San Diego Cancer Center, La Jolla, California
  - University of Chicago, Chicago, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - State University of New York Upstate Medical University, Syracuse, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Vermont, Burlington, Vermont